CLINICAL TRIAL: NCT06843174
Title: Perioperative Rectal Methadone in Spine Surgery
Acronym: PROMISE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: AFP Innovation Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: P-004
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Spinal Surgery; Post-operative Care; Post-operative Pain Management
Keywords: Intraoperative Methadone; Rectal Methadone administration; spinal surgery post-operative pain management

STUDY DESIGN:
Intervention Model Description: Randomized, placebo control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm with Methadone (Experimental): During the spinal surgery intervention, participants receive a single dose of 0.2mg/kg of Methadone rectally, after anesthesia induction.
  Interventions: Drug: Rectal Methadone administer during spinal surgery
- Placebo arm (Placebo Comparator): During the spinal surgery intervention, participants receive a single dose of saline solution rectally after anesthesia induction.
  Interventions: Other: Placebo: Rectal saline solution

INTERVENTIONS:
Drug: Rectal Methadone administer during spinal surgery — Rectal Methadone administered during spinal surgery for post-operative pain management
  Arms: Intervention Arm with Methadone
Other: Placebo: Rectal saline solution — Placebo: Rectal saline solution single dose received during surgery
  Arms: Placebo arm

SUMMARY:
Patients undergoing spinal surgery require pain control medication after their surgery. Investigators have successfully used intravenous Methadone to manage pain after surgery. However, doctors in Canada do not have the intravenous form of Methadone to prescribe to their patients. The investigators in Canada propose a pilot trial to investigate whether Methadone administered rectally could be used to manage pain after spinal surgery.

The main questions are:

1. Are investigators able to recruit participants for this trial and learn from this study to plan a larger trial?
2. Does Methadone administered rectally during surgery, reduce participants' pain intensity, use less pain medication, and have a better recovery after surgery? Investigators will compare Methadone to a placebo (a look-alike substance that contains no drug) to see if Methadone works to manage pain after surgery better than the usual pain management.

Participants will:

* receive either Methadone or placebo during surgery.
* be asked some questions about their pain during days 1 to 3 after surgery
* be contacted by phone to ask about their recovery

At this time, the study aims to recruit 40 participants from St. Michael's Hospital, to learn whether it will be feasible to plan a larger study.

DETAILED DESCRIPTION:
Indication: Adult patients undergoing spine surgery Condition: Perioperative pain management Number of participants 40 Primary outcome Feasibility (recruitment success, consent rate, adherence, patient withdrawal, missing data, adverse outcomes) Secondary outcome 1) Average pain intensity; 2) Rate of respiratory depression and postoperative ileus; 3) Use of opioids in morphine equivalents; 4) Quality of recovery Study design

* Interventional trial
* Allocation: Randomized
* Intervention model: 2-Arm Parallel-Group
* Primary purpose: Feasibility
* Phase: Phase IV

Masking Participants and Outcome Assessors

Study Intervention:

* Intervention Arm: Methadone 0.2mg/kg of ideal body weight via rectal administration + standard or care
* Placebo Arm: Saline solution via rectal administration + standard of care

Follow-Up: Postoperative days 1, 2, 3, and 30

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years-old.
2. Elective spinal surgery with fusion of one or more sacral, lumbar, thoracic, and/or cervical levels
3. Capacity to provide informed consent
4. For participants of childbearing potential, use of contraception.

Exclusion Criteria:

1. American Society of Anesthesiologists Physical Status > IV
2. Hypersensitivity to the active substance (methadone hydrochloride) or other opioid analgesics or to any ingredient in the formulation
3. Pregnant or nursing participants
4. Known or suspected mechanical gastrointestinal obstruction
5. Acute respiratory depression, elevated carbon dioxide levels in the blood, cor pulmonale, or pulmonary disease necessitating home oxygen therapy
6. Acute alcohol intoxication, delirium tremens, and convulsive disorders secondary to alcohol intoxication
7. Severe central nervous system depression, increased intracranial pressure, or head injury
8. Use of monoamine oxidase (MAO) inhibitors, such as isocarboxazid, phenelzine, selegiline, and tranylcypromine, within 14 days of enrollment
9. Diarrhea associated with pseudomembranous colitis caused by cephalosporins, lincomycins, or penicillins
10. Preoperative renal insufficiency or failure
11. Significant liver disease (cirrhosis or hepatic failure)
12. History of opioid use disorder within the last 3 months
13. Patients taking more than 90 mg of morphine equivalents daily
14. Poor comprehension of the English language
15. Patients who are likely to remain intubated postoperatively
16. QT interval > 500ms on preoperative ECG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility to recruit 40 participants into a trial of methadone and placebo | 18 months
  Recruitment rate (Acceptability and feasibility study)
Feasibility to recruit 40 participants into a trial of methadone and placebo | 18 months
  Withdrawal rate (Acceptability and feasibility study)

SECONDARY OUTCOMES:
Adverse outcomes | At 24, 48, and 72 hours post operative
  Rate of postoperative respiratory depression
Adverse outcomes | At 24, 48, and 72 hours post operative
  Rate of postoperative ileus
Opioid reduction | At 24, 48, and 72 hours post operative
  Total morphine equivalent used
Pain intensity after surgery | At 24, 48, and 72 hours post operative
  Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS) Pain Intensity, Pain intensity scale- 0 to 10 (The higher the number the higher the pain intensity)
Quality of Recovery | At 24, 48, and 72 hours post operative
  Quality of Recovery (QoR-15) Score, 15 items are rated on a 0-10 scale, with the total possible score ranging from 0 to 150, where higher scores indicate better recovery.
Pain interference | Difference between Baseline and 30 days after surgery
  Patient-Reported Outcomes Measurement Information System Pain Interference, PROMIS 6 a. 6 items, 5 Likert scale (the higher the score the higher the interference from pain)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Pereira, MD PhD, Principal Investigator — St. Michael's Hospital. Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a feasibility pilot trial only.

REFERENCES:
- [Background] Dale O, Sheffels P, Kharasch ED. Bioavailabilities of rectal and oral methadone in healthy subjects. Br J Clin Pharmacol. 2004 Aug;58(2):156-62. doi: 10.1111/j.1365-2125.2004.02116.x. PMID 15255797
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Deshur MA, Vender JS, Benson J, Newmark RL. Clinical Effectiveness and Safety of Intraoperative Methadone in Patients Undergoing Posterior Spinal Fusion Surgery: A Randomized, Double-blinded, Controlled Trial. Anesthesiology. 2017 May;126(5):822-833. doi: 10.1097/ALN.0000000000001609. PMID 28418966
- [Background] Machado FC, Vieira JE, de Orange FA, Ashmawi HA. Intraoperative Methadone Reduces Pain and Opioid Consumption in Acute Postoperative Pain: A Systematic Review and Meta-analysis. Anesth Analg. 2019 Dec;129(6):1723-1732. doi: 10.1213/ANE.0000000000004404. PMID 31743194
- [Background] Murphy GS, Avram MJ, Greenberg SB, Shear TD, Deshur MA, Dickerson D, Bilimoria S, Benson J, Maher CE, Trenk GJ, Teister KJ, Szokol JW. Postoperative Pain and Analgesic Requirements in the First Year after Intraoperative Methadone for Complex Spine and Cardiac Surgery. Anesthesiology. 2020 Feb;132(2):330-342. doi: 10.1097/ALN.0000000000003025. PMID 31939849
- [Background] Machado FC, Palmeira CCA, Torres JNL, Vieira JE, Ashmawi HA. Intraoperative use of methadone improves control of postoperative pain in morbidly obese patients: a randomized controlled study. J Pain Res. 2018 Oct 2;11:2123-2129. doi: 10.2147/JPR.S172235. eCollection 2018. PMID 30323647
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Elliott K, Kest B, Man A, Kao B, Inturrisi CE. N-methyl-D-aspartate (NMDA) receptors, mu and kappa opioid tolerance, and perspectives on new analgesic drug development. Neuropsychopharmacology. 1995 Dec;13(4):347-56. doi: 10.1016/0893-133X(95)00083-P. PMID 8747759
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Weir S, Samnaliev M, Kuo TC, Ni Choitir C, Tierney TS, Cumming D, Bruce J, Manca A, Taylor RS, Eldabe S. The incidence and healthcare costs of persistent postoperative pain following lumbar spine surgery in the UK: a cohort study using the Clinical Practice Research Datalink (CPRD) and Hospital Episode Statistics (HES). BMJ Open. 2017 Sep 11;7(9):e017585. doi: 10.1136/bmjopen-2017-017585. PMID 28893756
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Puvanesarajah V, Liauw JA, Lo SF, Lina IA, Witham TF, Gottschalk A. Analgesic therapy for major spine surgery. Neurosurg Rev. 2015 Jul;38(3):407-18; discussion 419. doi: 10.1007/s10143-015-0605-7. Epub 2015 Feb 14. PMID 25680636